CLINICAL TRIAL: NCT02500030
Title: Effects of Air Stacking Versus Glossopharyngeal Breathing on Maximum Insufflation Capacity in Children and Adolescents With Neuromuscular Disease
Brief Title: Air Stacking vs Glossopharyngeal Breathing in Neuromuscular Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Rodrigo Torres, Rodrigo Torres-Castro, University of Chile
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KIN2013-1
Record Dates: First submitted 2015-07-09; First posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Neuromuscular Diseases
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Air Stacking (Experimental): Air Stacking was performed with the subject seated in his wheelchair using a manual resuscitation bag (LIFESAVER® model 5345, Hudson, Temecula, USA) connected to a corrugated tube with an internal diameter of 22 mm, a one-way valve and a pipette. The maximum capacity of the bag was 1600 mL. A chest physiotherapist insufflated the patient during the inspiratory phase, requesting that inspire as much air as possible
  Interventions: Procedure: Air Stacking
- Glossopharyngeal Breathing (Experimental): Glossopharyngeal Breathing was also performed with the subject seated in his wheelchair and performing successive maneuvers of "swallowing air" until the maximum volume achieve was maintained. Then, the patient was instructed to breathe through ventilometer to register the MIC. Three measurements for each of the techniques were performed, and the highest reading was recorded. A difference of <10% between the measurements was used as the repeatability criterion
  Interventions: Procedure: Glossopharyngeal Breathing

INTERVENTIONS:
Procedure: Glossopharyngeal Breathing — Glossopharyngeal Breathing is a type of lung recruitment technique where the patients take a multiple inssuflations with their glossopharyngeal muscle.
  Arms: Glossopharyngeal Breathing
Procedure: Air Stacking — Air Stacking is a type of lung volume recruitment technique where insufflations are stacked in the lungs to maximally expand them, here done with a manual resuscitator.
  Arms: Air Stacking

SUMMARY:
Neuromuscular diseases (NMD) are characterized by a reduced maximum insufflation capacity (MIC), which contributes to increased morbidity and mortality from respiratory diseases. Techniques such as glossopharyngeal breathing (GPB) and insufflation using a manual resuscitation bag, or "air stacking (AS)", can be used to increase the MIC. These techniques employ different mechanisms, and the ability to learn the technique plays a key role in its proper implementation and effectiveness. The objective is compare the effects of AS and GPB on the MIC in patients with NMD.

Children and adolescents with NMD who were users of non-invasive mechanical ventilation were recruited. Vital capacity (VC) and MIC were measured prior to and after the intervention with AS and GPB. Values were compared pre- and post-intervention and were considered statistically significant if p <0.05.

DETAILED DESCRIPTION:
In neuromuscular diseases (NMD), progressive weakness of the respiratory muscles causes changes in the cough mechanism and prevents the elimination of secretions, which is the main cause of morbidity and mortality in this population.

Improving the cough response and achieving effective secretion elimination is required to increase lung volume and optimize the peak cough flow (PCF). It has been shown that a high PCF decreases respiratory complications in NMD. Vital capacity (VC) and maximum insufflation capacity (MIC) are the most important factors in increasing the PCF and, consequently, obtaining a more effective cough; thus, optimizing the lung volumes to achieve an adequate cough flow is important for effective bronchial hygiene. Currently, manual techniques are used to increase the MIC to achieve an effective PCF.

The most important manual techniques used to improve the MIC and, consequently the PCF, are air stacking (AS) and glossopharyngeal breathing (GPB). These have the advantages of low cost, patient autonomy and relative ease of learning compared to other techniques using electromechanical devices (e.g., volumetric ventilators and mechanical cough assist devices), whose main disadvantages are the high cost and complexity of use. AS involves delivering multiple breaths into a manual resuscitation bag and holding the insufflation volumes with the momentary closure of the glottis, which is repeated until the MIC is reached. GPB uses the glossopharyngeal muscles to successively introduce small amounts of air into the lungs to induce coughing and assist the weak inspiratory muscles. These techniques have been useful in treating different NMD, such as Spinal Muscular Atrophy (SMA) Type II, Duchenne Muscular Dystrophy (DMD) and Spinal Cord Injury (SCI).

The aim of this study was to compare the effects of two low-cost techniques, AS and GPB, on the MIC in children and adolescents with NMD. The hypothesis of this investigation was that although both techniques are effective, using AS results in a higher MIC than GPB.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of NMD
* Without respiratory exacerbation in the past 30 days
* No prior knowledge of the AS or GPB techniques
* Ability to understand instructions

Exclusion Criteria:

* Tracheostomized patients
* Incomplete glottis closure

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Vital Capacity | 30 minutes
  Vital Capacity is the volume of air expired after a maximal inspiration. The units are mililiters

SECONDARY OUTCOMES:
Peak Cough Flow | 30 minutes
  The peak cough flow is the maximal flow generated after a cough. The units of measure are Liters per minute

CONTACTS AND LOCATIONS:
Overall Officials: Homero Puppo, MSc, Principal Investigator — University of Chile